CLINICAL TRIAL: NCT05879328
Title: Liver Transplantation in Patients With Partial or Complete Response After Atezolizumab Plus Bevacizumab for Intermediate-advanced Stage Hepatocellular Carcinoma: the ImmunoXXL Study
Brief Title: The ImmunoXXL Study
Acronym: ImmunoXXL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Principal Investigator, Vincenzo Mazzaferro, Professor, MD, PhD, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Other Study IDs: INT 30/23
Record Dates: First submitted 2023-03-24; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver transplantation; Immune checkpoint inhibitors; Downstaging
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Immune profiling is performed (on day of transplantation, 3, 7, 15, 30, 90 days after transplantation with additional sampling at 6 months) by high resolution flow cytometry (Cytoflex platform) quantifying T cell effector and memory cell subsets (CD3, CD4 and others), T cell subsets associated with response to immunotherapy (PD1, CD28 and others), T reg cell subsets and myeloid cell subsets. Specific antiviral (HCV, HBV, EBV and CMV) and anti-tumor (HCC antigen pool including NY-Eso1, AFP and others) T cell activity is analyzed through ex-vivo peptide stimulation and specific IFNg release detected by Elispot. Immunomodulating and inflammatory cyto- and chemokines levels are quantified through secretome analysis (Cytokine Bead-Array o Fireplex). PBMC and plasma biobanking is performed as backup and for subsequent functional analysis (miRNA profiling,TCR repertoire and Rnaseq of blood immune cell subsets).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Liver Transplantation — Liver transplantation (LT) is an accepted surgical therapy for hepatocellular carcinoma (HCC) in patients who achieve effective and sustained tumor downstaging; in this study liver transplantation will be performed in patients undergoing a successful hepatocellular carcinoma (HCC) downstaging with the combination of atezolizumab and bevacizumab.

SUMMARY:
This study is aimed at confirming data of efficacy and safety of liver transplantation (LT) in patients with hepatocellular carcinoma (HCC) beyond current transplant criteria who demonstrate a sustained partial or complete radiological response to the atezolizumab and bevacizumab combination treatment, prescribed after completion of loco-regional therapies or as a first line systemic treatment.

The aim of the study is to demonstrate that liver transplantation, after effective HCC downstaging with atezolizumab and bevacizumab combination, may confer a survival benefit over atezolizumab and bevacizumab maintained treatment alone and that this strategy (tested in a consecutive non-randomized cohort) is not undermined by added risks.

DETAILED DESCRIPTION:
Liver transplantation (LT) is an accepted treatment for hepatocellular carcinoma (HCC). For patients with intermediate-advanced stage hepatocellular carcinoma (HCC) otherwise not eligible to curative treatments, tumor downstaging to LT is now an accepted strategy, as transplantation after a successful downstaging with loco-regional treatments confers a significant benefit in survival and recurrence/progression free survival compared to non-transplant strategies. Immune checkpoint inhibitors (ICIs) efficacy has been proven both as an adjuvant treatment in surgically treated HCCs and as a first line systemic therapy for advanced stage patients; in both cases with more than tolerable safety profiles. Therefore there is interest in using immunotherapy as a downstaging treatment prior to curative liver transplantation (LT).

This observational prospective single-arm study enrols patients on the transplant list after the achievement of a sustained radiological partial response (PR) or complete response (CR) on treatment with atezolizumab (flat dose of 1200 mg) and bevacizumab (15 mg/Kg) given intravenously every three weeks for a non otherwise treatable intermediate-advanced HCC.

Radiological response has to be sustained (for at least 3 months) and accompanied by a level of alpha fetoprotein (AFP) ≤ 100 UI/ml, if levels > 100 UI/ml at baseline or by decrease of the level of AFP parallel to the modified response evaluation criteria in solid tumors (mRECIST), if baseline levels ≤ 100 UI/ml.

Radiological and biochemical responses need to satisfy a ≥60% post-transplant survival at 5 years according to the Metroticket 2.0 calculator (www.hcc-olt-metroticket.org).

While on the liver transplant waiting list, treatment with atezolizumab and bevacizumab will be stopped. Treatment may be restored, according to clinical judgement:

* if waiting time on transplant list > 2 months
* if radiological and/or AFP progression within transplant criteria (predicted 5 year survival according to Metroticket 2.0 calculator ≥60%).
* if radiological and/or AFP progression beyond transplant criteria (predicted 5 year survival according to Metroticket 2.0 calculator < 60%); patients will be delisted (drop out) and treated according to clinical judgement and local standards.

Priority on the waiting list will follow local standards for candidates with HCC at risk of progression. Both donation after brain death (DBD) and after cardiac death (DCD) will be accepted for organ procurement.

Participants will also undergo a comprehensive blood immunomonitoring in order to explore the effect of liver transplantation and of related immunosuppressive regimens on the anti-tumoral immunomediated environment induced by the combination of atezolizumab and bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 and < 75 years
* signed Informed Consent Form
* hepatocellular carcinoma (HCC) previously diagnosed by histology/cytology or clinically by the American Association for the Study of Liver Disease (AASLD) criteria in cirrhotic patients. Patients without cirrhosis require compulsory histological confirmation of diagnosis.
* hepatocellular carcinoma (HCC) at diagnosis beyond "AFP-adjusted up-to-seven criteria" not amenable to loco-regional treatments and with sustained (at least 3 months) complete o partial response according to mRECIST after systemic treatment with atezolizumab and bevacizumab
* no major contraindications (cardiological, pulmonary, mental and social) to transplantation.

Exclusion Criteria:

* presence of extra-hepatic spread (EHS) defined as organ involvement other than the liver and hilar lymphnodes with short axis > 2 cm
* presence of tumoral portal vein thrombosis invading the main portal trunk for more than 1 cm in cranio-caudal extension (measured at coronal reconstructions scans at contrast enhanced CT/MRI).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intermediate-advanced HCC patients achieving complete response (CR) or partial response (PR) on treatment with atezolizumab and bevacizumab (approved dosages).
  Radiological response has to be sustained (for at least 3 months) and accompanied by a level of alpha fetoprotein (AFP) ≤ 100 UI/ml if levels > 100 UI/ml at baseline or by decrease of the level of AFP parallel to the mRECIST response, if baseline levels >100 UI/ml, to confirm a partial response (PR).
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | up to 2 years
  Recurrence-free survival (RFS) is defined as the interval (in months) between the date of transplantation and the date on which tumor recurrence is detected at any site at contrast-enhanced computed tomography (CT) or magnetic resonance imaging (MRI) scan, calculated in the entire collected patient population with censoring at the date of death or last follow-up in recurrence-free patients

SECONDARY OUTCOMES:
Tumor response | From the time of signature of informed consent until the date of first documented progression or date of death from any cause, whichever comes first, assessed up to 48 months
  Tumor response at radiology (contrast enhanced CT scan or MRI) is defined as overall response rate (ORR) that is the number of radiological responses divided by the number of patients:
  * complete response (CR) is defined by the disappearance of any arterial enhancement in all target lesions according to mRECIST criteria
  * partial response (PR) is defined by ≥50% decrease in the sum of diameters of viable target lesions, taking as reference the baseline sum of the diameters of target lesions
  Pathological response at histology is assessed as the percentage of surface with non-viable cancer cells (represented by necrosis or fibrosis) in relation to the total tumor area and is equal to: 100% - viable cancer cells (%). If there are multiple tumors, the mean percentage is used. Complete pathological response (pCR) is defined by the absence of viable tumor cells in any nodule
Complication rate | monthly, up to 2 years
  Complication rate is defined as the number of complications, deviating from the normal post-operative course, divided by the number of patients; complications will be assessed according to Dindo-Clavien classification. The total number of both transplant-related and treatment-related adverse events (graft failure, histology confirmed acute rejection, hospital-treated infections) assessed by the Common Terminology Criteria for Adverse Events (CTCAE) v.4.0 will also be divided by the number of participants
Overall survival (OS) | up to 2 years
  Overall survival (OS) is defined as the interval (in months) between the date of transplantation and the date of death for any reason in the entire collected patient population, with censoring at the date of last follow-up in alive patients
Patients' reported outcomes (PROs) | every 3 months for the first six months, then every 6 months up to 2 years
  Patients' reported outcomes will be evaluated by the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC QLQ-C30, version 3) filled in by all participants in order to measure health related quality of life.
  The QLQ-C30 is composed of 28 multi-item scales rated from 1 to 4 (where 1 is "not at all", 2 is "a little", 3 is "quite a bit" and 4 is "very much") and 2 single-item measures rated from 1 to 7, where 1 is "very poor" and 7 is "excellent". These items include five functional scales, three symptom scales, a global health status scale, and six single items. The scales produce a final score ranging from 0 to 100. A high scale score represents a higher response level. In detail:
  * a high score for a functional scale represents a high / healthy level of functioning
  * a high score for the global health status represents a high QoL
  * a high score for a symptom scale / item represents a high level of symptomatic problems
Comparison with historical series | up to 2 years
  As this study has no comparator arm, overall survival (OS) and recurrence free survival (RFS) of the participants to the study will be compared with the overall survival (OS) and recurrence free survival (RFS) of historical series of patients with intermediate-advanced HCC downstaged using loco-regional treatments only (doi:10.1016/S1470-2045(20)30224-2, PMID 32615109) and of patients treated with and responding to atezolizumab and bevacizumab in the advanced tumor setting (doi:10.1056/NEJMoa1915745, PMID: 32402160)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Mazzaferro, MD, PhD, Principal Investigator — Fondazione Istituto Nazionale Tumori Milano - Italy
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mazzaferro V, Citterio D, Bhoori S, Bongini M, Miceli R, De Carlis L, Colledan M, Salizzoni M, Romagnoli R, Antonelli B, Vivarelli M, Tisone G, Rossi M, Gruttadauria S, Di Sandro S, De Carlis R, Luca MG, De Giorgio M, Mirabella S, Belli L, Fagiuoli S, Martini S, Iavarone M, Svegliati Baroni G, Angelico M, Ginanni Corradini S, Volpes R, Mariani L, Regalia E, Flores M, Droz Dit Busset M, Sposito C. Liver transplantation in hepatocellular carcinoma after tumour downstaging (XXL): a randomised, controlled, phase 2b/3 trial. Lancet Oncol. 2020 Jul;21(7):947-956. doi: 10.1016/S1470-2045(20)30224-2. PMID 32615109
- [Background] Reig M, Forner A, Rimola J, Ferrer-Fabrega J, Burrel M, Garcia-Criado A, Kelley RK, Galle PR, Mazzaferro V, Salem R, Sangro B, Singal AG, Vogel A, Fuster J, Ayuso C, Bruix J. BCLC strategy for prognosis prediction and treatment recommendation: The 2022 update. J Hepatol. 2022 Mar;76(3):681-693. doi: 10.1016/j.jhep.2021.11.018. Epub 2021 Nov 19. PMID 34801630
- [Background] Llovet JM, Castet F, Heikenwalder M, Maini MK, Mazzaferro V, Pinato DJ, Pikarsky E, Zhu AX, Finn RS. Immunotherapies for hepatocellular carcinoma. Nat Rev Clin Oncol. 2022 Mar;19(3):151-172. doi: 10.1038/s41571-021-00573-2. Epub 2021 Nov 11. PMID 34764464
- [Background] Finn RS, Qin S, Ikeda M, Galle PR, Ducreux M, Kim TY, Kudo M, Breder V, Merle P, Kaseb AO, Li D, Verret W, Xu DZ, Hernandez S, Liu J, Huang C, Mulla S, Wang Y, Lim HY, Zhu AX, Cheng AL; IMbrave150 Investigators. Atezolizumab plus Bevacizumab in Unresectable Hepatocellular Carcinoma. N Engl J Med. 2020 May 14;382(20):1894-1905. doi: 10.1056/NEJMoa1915745. PMID 32402160
- [Background] Mazzaferro V, Sposito C, Zhou J, Pinna AD, De Carlis L, Fan J, Cescon M, Di Sandro S, Yi-Feng H, Lauterio A, Bongini M, Cucchetti A. Metroticket 2.0 Model for Analysis of Competing Risks of Death After Liver Transplantation for Hepatocellular Carcinoma. Gastroenterology. 2018 Jan;154(1):128-139. doi: 10.1053/j.gastro.2017.09.025. Epub 2017 Oct 5. PMID 28989060
- [Background] Hack SP, Spahn J, Chen M, Cheng AL, Kaseb A, Kudo M, Lee HC, Yopp A, Chow P, Qin S. IMbrave 050: a Phase III trial of atezolizumab plus bevacizumab in high-risk hepatocellular carcinoma after curative resection or ablation. Future Oncol. 2020 May;16(15):975-989. doi: 10.2217/fon-2020-0162. Epub 2020 Apr 30. PMID 32352320
- See also: Survival prognosis calculator in patients with HCC undergoing liver transplantation — http://www.hcc-olt-metroticket.org/